CLINICAL TRIAL: NCT02276352
Title: An Open, Randomized, Three-way Cross-over Study in Healthy Volunteers to Evaluate the Relative Bioavailability of Meloxicam After Single p.o. Administration of 2 x 7.5 mg Meloxicam Tablets Compared to 15 mg Meloxicam Tablet, and Dose-proportionality Over a Dosage Range of 7.5 mg and 15 mg.
Brief Title: Relative Bioavailability of Meloxicam 2 x 7.5 mg Tablets Compared to 15 mg Tablet and Dose Proportionality Over a Dose Range of 7.5 mg and 15 mg in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.226
Record Dates: First submitted 2014-10-27; First posted 2014-10-28 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-05

CONDITIONS: Healthy

ARMS (3):
- Meloxicam low dose - one tablet (Experimental)
  Interventions: Drug: Treatment 1
- Meloxicam high dose - two tablets (Experimental)
  Interventions: Drug: Treatment 2
- Meloxicam high dose - one tablet (Active Comparator)
  Interventions: Drug: Treatment 3

INTERVENTIONS:
Drug: Treatment 1
  Arms: Meloxicam low dose - one tablet
Drug: Treatment 2
  Arms: Meloxicam high dose - two tablets
Drug: Treatment 3
  Arms: Meloxicam high dose - one tablet

SUMMARY:
Study to assess the relative bioavailability of two 7.5 mg meloxicam tablets (American type) compared to one 15 mg meloxicam tablet (American type), and to investigate dose-proportionality over the dosage range 7.5 mg to 15 mg

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age >= 18 and <= 50 years
* Broca >= -20% and <= + 20 %

Exclusion Criteria:

* Any finding of the medical examination (including laboratory blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastro-intestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* Hypersensitivity to meloxicam and/or non-steroidal antirheumatic agents
* Intake of drugs with a long half-life (>24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smoker (>= 10 cigarettes or >= 3 cigars or >= 3 pipes/day)
* Inability to refrain from smoking on study days
* Alcohol abuse
* Drug abuse
* Blood donation (<= 1 months prior to administration)
* Excessive physical activities (<= 5 days prior to administration)
* History of hemorrhagic diatheses
* History of gastro-intestinal ulcer, perforation or bleeding
* History of bronchial asthma

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. sterilization, intrauterine device (IUD), oral contraceptives
* Inability to maintain this adequate contraception during the whole study period
* Lactating

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1999-06; Primary Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose

SECONDARY OUTCOMES:
Time from dosing to the maximum concentration of the analyte in plasma (tmax) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Total area under the plasma drug concentration time curve (AUC) from time of administration to the time of the last quantifiable drug concentration (AUC0-t) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Apparent terminal elimination rate constant (λz ) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Terminal half-life of the analyte in plasma (t½) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Mean residence time (MRTtot) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Apparent volume of distribution of the analyte during the terminal phase (Vz/F) | predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 14, 24, 32, 48, 72 and 96 hours postdose
Number of patients with abnormal findings in pulse rate | predose, up to 96:00 h post dose
Number of patients with abnormal findings in systolic and diastolic blood pressure | predose, up to 96:00 h post dose
Number of patients with adverse events | up to 39 days
Number of patients with abnormal changes in laboratory parameters | predose, up to 96:00 h post dose